CLINICAL TRIAL: NCT01273012
Title: Cost-effectiveness of Infloran (TM) in Treating Acute Childhood Diarrhea in Phramongkutklao Hospital
Acronym: infloran
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: LTC Nopaorn Phavichitr, Department of Pediatrics, Phramongkutklao Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: P001h/53
Record Dates: First submitted 2011-01-03; First posted 2011-01-10 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Acute Diarrhea
Keywords: probiotic; cost-effectiveness; diarrhea; children; Sum of the monetary cost of the hospitalization
MeSH Terms: conditions — Diarrhea | interventions — acidocin D20079, Lactobacillus acidophilus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The group of patients treated with placebo.
  Interventions: Drug: Probiotic - Infloran
- Infloran (Experimental): The group of patients treated with Infloran.
  Interventions: Drug: Probiotic - Infloran

INTERVENTIONS:
Drug: Probiotic - Infloran — Drug:Probiotic - Infloran (TM) 1 cap (1 billion CFU of L. acidophilus and 1 billion CFU of B. bifidum) PO bid or tid
  Other Names: Infloran; L. acidophilus; B. bifidum

SUMMARY:
The purpose of this study is to determine whether the probiotic Infloran is cost-effective in treating acute childhood diarrhea.

DETAILED DESCRIPTION:
Probiotics have been proved to shorten duration of diarrhea in children; whether they are cost-effective is less clear. We'd like to validate the use of Infloran, a proprietary probiotic sold in Thailand, in terms of its cost-effectiveness compared to standard diarrhea care in our hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Children 3 months to 6 years of age
* Hospitalized due to acute diarrhea

Exclusion Criteria:

* History of probiotic treatment in this episode of illness
* History of use of other anti-diarrheal medications
* Chronic gastrointestinal disease(s)
* Severe dehydration
* Severe systemic disease(s)

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
monetary cost of hospitalization in Thai Baht | from admission to discharge date, approximately 1-7 days

SECONDARY OUTCOMES:
days of hospitalization | from admission to discharge date, approximately 1-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Nopaorn Phavichitr, MD, Principal Investigator — Department of Pediatrics, Phramongkutklao
Locations (1):
- Department of Pediatrics, Phramongkutklao Hospital, Bangkok, Thailand